CLINICAL TRIAL: NCT00156442
Title: OSAS in Children With Cleft Lip/Palate
Brief Title: A Study to Examine the Relationship Between Sleep Apnea and Cleft Lip/Palate
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: John Girrotto MD, U of Rochester
Other Study IDs: 11595
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2006-09

CONDITIONS: Obstructive Sleep Apnea Syndrome; Cleft Lip/Palate
Keywords: Obstructive Sleep Apnea Syndrome; Cleft lip/palate; Children
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study is to examine the relationship between sleep apnea and neurocognitive behaviors in children with cleft lip/palate. Describe the incidence and severity of obstructive sleep apnea in an unselected population of grade school aged children with surgically repaired cleft palate.

A. Is the incidence of OSA higher in children with cleft palate than age matched historical control groups? B. Are nighttime symptoms an adequate screening tool to exclude the diagnosis of OSA in children with surgically repaired cleft palate? Describe the velopharyngeal closure patterns during speech in an unselected population of grade school aged children with surgically repaired cleft palate. Describe the neurobehavioral phenotype of an unselected population of grade school aged children with surgically repaired cleft palate.

DETAILED DESCRIPTION:
Obstructive sleep apnea is closely associated with measurable, impaired cognitive function among otherwise neurologically normal, healthy children . In addition, at least one recent study has reported mild hyperactive-impulsive symptoms among children with sleep disordered breathing . Cleft lip and cleft palate comprise the fourth most common birth defect affecting 1 in 700 newborns. Despite surgical repair, nearly one in four children with surgically repaired cleft palate will have significant velopharyngeal dysfunction . Velopharyngeal closure is expected in nearly all sounds in the English language. As a result, incompetence results in significant speech disability. Because hypernasal speech patterns are more functionally disabling than hyponasality, surgeons tend to err on the side of over-closure of the nasopharynx in an effort to improve the intelligibility of a child's speech when performing secondary speech procedures. Thus, surgical speech procedures are well known to result in clinically significant obstructive sleep apnea . Unfortunately, no data exists about the impact of obstructive sleep apnea on neurocognitive function in children with cleft palate raising the possibility that surgical intervention aimed at improving speech may result in neurocognitive disabilities due to obstructive sleep apnea. Furthermore, no data exists to guide surgeons as to the relative impact of poor speech versus sleep apnea on global neurocognitive and academic functioning. We therefore hypothesize that unrecognized obstructive sleep apnea occurs in patients with surgically repaired cleft palate and results in demonstrable neurobehavioral sequelae. In order to address these hypotheses, we propose the following specific aims:

Specific Aim #1:

Describe the incidence and severity of obstructive sleep apnea in an unselected population of grade school aged children with surgically repaired cleft palate.

A. Is the incidence of OSA higher in children with cleft palate than age matched historical control groups? B. Are nighttime symptoms an adequate screening tool to exclude the diagnosis of OSA in children with surgically repaired cleft palate? Detailed measurement of respiratory disturbances during sleep affecting both gas exchange and sleep state continuity will be performed via polysomnography. Comparisons will be made between snoring and non-snoring groups. Additional comparisons will be made with the literature where appropriate. Although sleep disordered breathing is well known to occur with increased frequency in children with craniofacial anomalies, the specific incidence in children with cleft palate remains unknown. Whether snoring proves to be an adequate screening tool in children with cleft palate also remains to be proven. We hypothesize that sleep apnea affecting both gas exchange and sleep state continuity will be identified both in the presence and absence of habitual snoring.

Specific Aim #2:

Describe the velopharyngeal closure patterns during speech in an unselected population of grade school aged children with surgically repaired cleft palate. Detailed measurement of nasal acoustic energy while reading defined passages will be performed. Measured nasalance will be compared to assessment by a trained speech pathologist. Presence of substitutions of consonants valved at the level of the glottis or oral pharynx, a common feature of the misarticulations that develop when speech is acquired in the presence of velopharyngeal dysfunction will be noted. In keeping with published literature , we hypothesize that measured nasometry will correlate closely with speech pathologist assessment of nasality. Furthermore, we hypothesize that misarticulations will be noted more prominently in those children with velopharyngeal dysfunction.

Specific Aim #3:

Describe the neurobehavioral phenotype of an unselected population of grade school aged children with surgically repaired cleft palate. Detailed assessment of neurobehavior will be performed using the Behavior Rating Inventory of Executive Function (BRIEF), Parent & Teacher Forms and the Conners' Parent Rating Scale-Revised/Conners' Teacher Rating Scale (CPRS/CTRS). These questionnaires, which specifically test for executive function and behavioral/emotional problems respectively, are selected because these are the behaviors thought to be most affected by OSA. Comparisons will be made with normative data from the literature where appropriate. Cleft palate carries significant long-term medical, dental, educational and psychological burdens for those affected. We therefore hypothesize that significant neurobehavioral abnormalities will be identified in children with surgically repaired cleft palate

ELIGIBILITY:
Inclusion Criteria:

* 100 children with cleft lip/palate and signs and symptoms of OSAS, parents who can read and write English

Exclusion Criteria:

* Parents who cannot read and write English, children with severe neurological compromise

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children with celft palate and symptoms of OSA
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2005-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Girotto, MD, Principal Investigator — University of Rochester; Heidi V. Connolly, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States